CLINICAL TRIAL: NCT00028288
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Daclizumab in Patients With Chronic, Persistent Asthma
Brief Title: Study of Daclizumab in Patients With Chronic, Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAC-1003
Record Dates: First submitted 2001-12-19; First posted 2001-12-20 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Asthma
Keywords: Asthma; Daclizumab; anti-Tac monoclonal antibody; anti-IL-2; Zenapax
MeSH Terms: conditions — Asthma | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
The purpose of the study is to evaluate an investigational medication to treat chronic persistent asthma. The research is being conducted at up to 22 clinical research sites in the US and is open to both men and women ages 18 to 70 years old. Participants in the study will have a number of visits to a research site over a 10-month period. All study-related care and medication is provided to qualified participants at no cost: this includes all visits, examinations and laboratory work.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma for 6 or more months
* History of chronic persistent asthma requiring daily high dose inhaled corticosteroid for 3 or more months prior to enrollment

Exclusion Criteria:

* Patients with 10 or more pack years of smoking history or smoking within 12 months of study enrollment
* No significant disease other than asthma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2001-09; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Medical Research Associates, Long Beach, California
  - Southern California Research, Mission Viejo, California
  - Institute of Health Care Assessment, Inc., San Diego, California
  - Bensch Research Associates, Stockton, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Clinical Reserch Centers of Colorado, Denver, Colorado
  - Florida Center for Allergy and Asthma Reserch, Miami, Florida
  - Rx Research, Woodstock, Georgia
  - ICSL Clinical Studies, Bloomington, Illinois
  - Asthma and Allergy Center of Chicago, S.C., River Forest, Illinois
  - New England Clinical Studies, North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Princeton Center for Clinical Research, Princeton, New Jersey
  - Allergy, Asthma, and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Valley Clinical Research Center, Easton, Pennsylvania
  - Pharmaceutical Research and Consulting, Inc., Dallas, Texas
  - University of Wisconsin Medical School, Madison, Wisconsin
  - Allergy and Respiratory Care Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Busse WW, Israel E, Nelson HS, Baker JW, Charous BL, Young DY, Vexler V, Shames RS; Daclizumab Asthma Study Group. Daclizumab improves asthma control in patients with moderate to severe persistent asthma: a randomized, controlled trial. Am J Respir Crit Care Med. 2008 Nov 15;178(10):1002-8. doi: 10.1164/rccm.200708-1200OC. Epub 2008 Sep 11. PMID 18787222